CLINICAL TRIAL: NCT04505579
Title: The Tether™ - Vertebral Body Tethering System Post Approval Study
Status: Recruiting | Type: Observational
Sponsor: ZimVie (Industry)
Collaborators: Setting Scoliosis Straight Foundation (Other); Exponent, Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: RAU2019-40S
Record Dates: First submitted 2020-07-20; First posted 2020-08-10 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Scoliosis Idiopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Tether: Patients who have received The Tether HUD for treatment of idiopathic scoliosis.
  Interventions: Device: Anterior Vertebral Body Tethering

INTERVENTIONS:
Device: Anterior Vertebral Body Tethering — Anterior Vertebral Body Tethering (AVBT) is a technique that utilizes growth modulation to remodel the shape of the vertebra and straighten scoliotic curves in skeletally immature individuals. In this technique, screws are inserted at each vertebral level for the length of the convex side of the curve. A strong cord is connected through the screw tulip heads and used to initially straighten the curve as each level is fixed with a set screw. Following surgery and during the growth period the spine begins to remodel according to the Hueter-Volkmann Law, bone growth is relatively inhibited in areas of increased pressure (convex or tethered side) and relatively stimulated in areas of decreased pressure or tension (concave side).
  Other Names: AVBT

SUMMARY:
This study is an opportunity to provide continued reasonable assurance of the safety and probable benefit of The Tether HUD. The study will collect long term safety and efficacy information from patients who have had their idiopathic scoliosis treated via anterior vertebral body tethering (AVBT) with The Tether.

DETAILED DESCRIPTION:
While spinal fusion remains the standard surgical treatment for progressive idiopathic scoliosis, concerns about the long-term effects of spinal fusion have led to the investigation of growth-modulation techniques. Anterior Vertebral Body Tethering (AVBT) is one such technique that utilizes growth modulation to remodel the shape of the vertebra and straighten scoliotic curves in skeletally immature individuals. In this technique, screws are inserted at each vertebral level for the length of the convex side of the curve. A strong cord is connected through the screw tulip heads and used to initially straighten the curve as each level is fixed with a set screw. Following surgery and during the growth period the spine begins to remodel according to the Hueter-Volkmann Law, bone growth is relatively inhibited in areas of increased pressure (convex or tethered side) and relatively stimulated in areas of decreased pressure or tension (concave side). Following this principle, AVBT has been shown to alter spinal growth with the potential to correct scoliosis while maintaining spine flexibility.

The objective of the study is to assess the ongoing safety and probable benefit of The Tether HUD which was approved by the FDA under an HDE. Subject enrollment and data collection will be managed by the Harms Study Group (HSG) and Setting Scoliosis Straight Foundation (SSSF) Registry. Institutions that are HSG members or affiliates, with Investigators/surgeons that are trained and approved to perform surgeries with The Tether, will participate in the registry. Ten sites from this group will be identified as study sites specific to this Tether post-approval study (PAS). Consecutive subjects from these sites, that meet the eligibility criteria of this study, will be flagged in the registry as the PAS cohort and the study endpoints will be assessed across this population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of progressive idiopathic scoliosis
* Skeletally immature, based on both Risser (<5) and Sanders (<8) assessments
* Major Cobb angle ≥30° and ≤65°
* Osseous structure dimensionally adequate to accommodate screw fixation, as determined by radiographic imaging
* Failed or intolerant to bracing

Exclusion Criteria:

* Presence of any systemic infection, local infection, or skin compromise at the surgical site
* Prior spinal surgery at the level(s) to be treated
* Documented poor bone quality, defined as a T-score -1.5 or less
* Any other medical or surgical condition which would preclude the potential benefit of spinal surgery, such as coagulation disorders, allergies to the implant materials, and patient's unwillingness or inability to cooperate with post-operative care instructions
* Unwillingness, inability, or living situation (e.g. custody arrangements, homelessness, detention) that would preclude ability to return to the study site for follow-up visits as described in protocol and Informed Consent
* Unwillingness to sign Informed Consent Form and participate in study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Tether™ - Vertebral Body Tethering System is indicated for skeletally immature patients that require surgical treatment to obtain and maintain correction of progressive idiopathic scoliosis, with a major Cobb angle of 30 to 65 degrees whose osseous structure is dimensionally adequate to accommodate screw fixation, as determined by radiographic imaging. Patients should have failed bracing and/or be intolerant to brace wear.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of SAEs and device- &/or procedure-related AEs | AVBT surgery to five year post-op
  The primary safety endpoint is the rate of Serious Adverse Events (SAEs) and device- and/or procedure-related Adverse Events (AEs)
Percentage of subjects with maintenance of the major Cobb angle less than or equal to 40 degrees at 60 months post-surgery | AVBT surgery to five year post-op
  The primary probable benefit endpoint is the percentage of patients with maintenance of the major Cobb angle less than or equal to 40 degrees at 60 months post-surgery

SECONDARY OUTCOMES:
Adverse Events | AVBT surgery to five year post-op
  Rates of overall Adverse Events; relatedness, severity, time to event
Reoperation | AVBT surgery to five year post-op
  Rates and types of reoperation
Number of participants with new curves that develop above or below the tethered portion of the spine. | AVBT surgery to five year post-op
  Determined by radiographic assessment, defined as a new curve development with Cobb angle measurement greater than or equal to 40 degrees.
Number of participants with secondary curves that progress to the point of clinical significance. | AVBT surgery to five year post-op
  Determined by radiographic assessment, typically defined as an increase in secondary Cobb angle measurement greater than or equal to 10 degrees, or medical intervention/ intent to treat.
Number of participants with device integrity failures including cord breakage and screw migration. | AVBT surgery to five year post-op
Mean (SD) and distributions of sagittal balance (mm) from pre-op through last visit | Baseline to five year post-op
  Sagittal balance is assessed on the lateral radiograph by measuring the difference (i.e. distance) between posterosuperior aspect of the S1 vertebral body and the plumb line.
Mean (SD) and distributions of lumbar lordosis (degrees) from pre-op through last visit. | Baseline to five year post-op
  Lumbar lordosis is defined as the angle at the intersection of lines perpendicular to lines parallel to the superior endplate of T12 and the superior endplate of S1.
Mean score of Scoliosis Research Society 22r Patient Questionnaire | Baseline to five year post-op
  Self-reported outcomes of function, pain, self-image, mental health, and satisfaction. Mean score; 5 (Best) - 1 (Worst)
Number of participants with compromised lung function | Baseline to five year post-op
  Comparison of the measured lung function (forced expiratory volume (FEV1), forced vital capacity (FVC) and FEV1/FVC) to predicted values, lower and upper limits of normal to determine if lung function is within the limits of the normal population.
Measurement (degrees rotation) of trunk shape by scoliometer device. Mean (SD) [min, max] will be reported. | Baseline to five year post-op
  Measurements of trunk shape or rib hump will be collected preoperatively and at each follow-up visit. A standard scoliometer device will be used to measure the rib hump in the thoracic and/or lumbar regions of the spine, as applicable. The scoliometer is laid across the curve at right angles with the 0° mark at the spinous process and resting gently on the skin, not pressed down. The degrees of rotation are read and recorded.
Trunk flexibility as determined by distance (cm) of flexion and lateral bend using fingertip to floor method. | Baseline to five year post-op

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Health, Jacksonville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ochsner Health, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri - Columbia, Columbia, Missouri
  - Mount Sinai, New York, New York
  - Shriners Children's Hopital, Philadelphia, Pennsylvania
  - Seattle Children's, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided